CLINICAL TRIAL: NCT00827281
Title: D-Cycloserine Enhancement of Exposure-Based CBT for Smoking Cessation
Brief Title: D-Cycloserine Enhancement of Exposure-Based CBT for Smoking Cessation (DCSSmoking)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not funded and pilot work proved impractical.
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Ph.D., Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1728
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Smokers
Keywords: DCS; CBT; smoking; tobacco
MeSH Terms: conditions — Smoking | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DCS-augmented CBT for smoking cessation
  Interventions: Drug: D-cycloserine
- 2 (Placebo Comparator): Placebo-augmented CBT for smoking cessation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — Single dosage prior to sessions 3, 4 & 5
  Other Names: DCS
  Arms: 1
Drug: Placebo — Single dosage prior to sessions 3, 4 & 5
  Arms: 2

SUMMARY:
This study examines whether isolated doses of D-cycloserine enhance the efficacy of CBT for smoking cessation.

DETAILED DESCRIPTION:
In comparison to placebo-augmented cognitive behavioral therapy (CBT), D-cycloserine-augmented CBT will lead to a greater reduction in both short-and long-term point prevalence abstinence as well as time to first smoking lapse and time to smoking relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Be a regular smoker for at least one year 3. Currently smoke an average of at least 10 cigarettes per day 4. Report a motivation to quit smoking in the next month of at least 5 on a 10 point scale 5. Score 20 or greater on the 16-item Anxiety Sensitivity Index (Schmidt & Joiner, 2002).

Exclusion Criteria:

1. Current diagnosis of a psychotic, eating, developmental or bipolar disorder (as determined by the SCID)
2. Current anxiety or mood disorder rated moderate or greater (i.e., CGI score of 4 or greater for an anxiety or depressive disorder or any current or recent-1 year--suicidal ideation)
3. Psychoactive substance abuse or dependence (excluding nicotine dependence) within the past 6 months
4. Current use of isoniazid psychotropic medication
5. A history of significant medical condition, such as cardiovascular, neurologic, gastrointestinal, pregnancy and/or breast feeding, history of seizure (other than febrile seizures in childhood) or other systemic illness and/or be deemed as currently unhealthy in the context of a complete physical examination
6. Limited mental competency and the inability to give informed, voluntary, written consent to participate,
7. Current use of any pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers during the quit attempt,
8. Concurrent psychotherapy initiated within three months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of anxiety or mood disorder other than general supportive therapy initiated at least 3 months prior to the study
9. Use of other tobacco products
10. Planning on moving (outside of the immediate area) in the next six months
11. Insufficient command of the English language (i.e., they cannot carry on a conversation with an interviewer in the English language or read associated text).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Carbon monoxide analysis | Baseline, Weeks 4, 5, 6, 7, 8, 9, 13, 21, & 29
Cotinine levels in saliva | Baseline, Weeks 21 & 29

SECONDARY OUTCOMES:
Anxiety Sensitivity Index | Baseline, Weeks 5, 6, 7, 8, 9, 13, 21 & 29
Minnesota Withdrawal Scale | Each visit
Mood & Anxiety Symptom Questionnaire | Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, & 8
Smoking Cessation Self-Efficacy | Baseline, Weeks 3, 4, 5, 6, 7, 8, 9, 13, 21 & 29

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States